CLINICAL TRIAL: NCT04207424
Title: EMbolisation Bariatrique de l'ARcade Gastro-épiploïque Chez Les Patients Obèses
Brief Title: Embolization of Arterial Gastric Supply in Obesity
Acronym: Embargo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients were selected but their very condition and the resulting comorbidities did not allow their inclusion. In addition, the health crisis prevented any bariatric operation of this complexity for an indefinite period.
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-005
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Morbid Obesity
Keywords: Bariatric embolization; Obesity; Metabolic syndrome
MeSH Terms: conditions — Obesity, Morbid; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization (Experimental): Patients undergoing embolization of the gastro-epiploic arcade
  Interventions: Procedure: Emblization of the gastro-epiploic arcade

INTERVENTIONS:
Procedure: Emblization of the gastro-epiploic arcade — Endovascular embolization of the gastro-epiploic arcade using 300-500 micrometres calibrated polyvinyl-alcohol microparticles

SUMMARY:
This study aims to assess safety and efficacy of bariatric embolization of the gastro-epiploic arcade using 300-500 micrometres calibrated polyvinyl-alcohol microparticles, for patients with morbid obesity.

DETAILED DESCRIPTION:
Obesity is now an epidemic in the developed and developing world. Medical management is ineffective at population level. Metabolic surgery has been shown to be effective in achieving weight loss and controlling associated conditions. However, surgery is invasive and has associated complications. Furthermore, not every patient is interested in or eligible for surgery.

Bariatric gastric embolization recently emerged as a promising minimally invasive alternative to open bariatric surgery. Data from several initial pilot clinical trials suggests that gastric embolization is safe and can induce weight loss.

Previous studies have concentrated on left gastric artery embolization as the primary target vessel because it supplies the largest portion of the fundus. However, it may be desirable to target a different artery, specifically the left gastroepiploic which also supplies the fundus. The left gastric artery is spared in bariatric surgery because it supplies the residual pouch after the surgery. Embolization of the left gastric artery may result in worse healing in the event of follow-up surgery potentially excluding people should they subsequently want it or become eligible.

This study aims to assess safety and efficacy of bariatric embolization of the gastro-epiploic arcade using 300-500 micrometres calibrated polyvinyl-alcohol microparticles, for patients with morbid obesity.

The target population consists of adult, morbidly obese patients with contraindication for bariatric surgery. Patients included in the study will be followed up for 12 months post bariatric embolization. The primary end point is procedural safety, defined as number and severity of adverse events occurring during the study period. Secondary end points include weight loss, evolution of weight and thigh circumferences, evolution of serum ghrelin levels and evolution of quality of life indexes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥18 and ≤ 71 years old
* BMI ≥ 40 or BMI ≥ 35 in association with one of the following comorbidities: hypertension, type 2 diabetes, obstructive sleep apnea
* Relative contraindication to bariatric surgery
* Able to sign informed consent.

Exclusion Criteria:

General

* Impossible or unwilling to attend follow-up visits.
* Weight > 250kg (weight limit of angiography table)
* Confirmed allergy to intravenous contrast agents.
* Pregnancy, breast feeding or willingness to conceive during the following year
* Impossible to maintain dorsal decubitus during intervention
* Life expectancy < 1 year
* Current enrollment in another clinical trial
* Arterial anatomy rendering embolization very difficult or impossible (as evaluated by investigators)
* Patient under the protection of justice
* Patient under guardianship or trusteeship

Gastro-intestinal

* Pre-existing chronic abdominal pain
* History of inflammatory bowel disease
* History of gastroparesis
* History of gastric surgery, gastric embolization or radiotherapy
* History of peptic ulcer
* Significant risk factors for peptic ulcer, including daily use of non-steroidal anti-inflammatory drugs, active smoking or active infection with Helicobacter pylori
* Abnormal upper digestive endoscopy

Hepatic

* Cirrhosis
* Portal venous hypertension
* Bilirubin > 2,0 mg/dL
* Albumin < 2,5 g/L

Cardiovascular

* Known aortic pathology i.e. aneurysm or dissection
* Severe peripheral arterial disease

Renal

- Renal failure, Creatinine Clearance < 60ml/min/1,73 m2

Hematologic/Immunologic/Oncologic/Infectious

* Acute or chronic infection
* Active cancer
* Auto-immune disease requiring immunosuppression
* Neutrophil count < 1,5 x 10 ^ 9/L
* Platelet count < 100 x 10 ^ 9/L

Contraindication to contrast medium Visipaque solution for injection

* Hypersensitivity to the active substance (Iodixanol) or to any of the excipients
* History of immediate major or delayed skin reaction to the injection of the product
* Decompensated heart failure
* Thyrotoxicosis
* Contraindication to the use of the embogold microsphere

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 7 days post embolization
Number of participants with adverse events | 1 month post embolization
Number of participants with adverse events | 3 months post embolization
Number of participants with adverse events | 6 months post embolization
Number of participants with adverse events | 12 months post embolization

SECONDARY OUTCOMES:
Change in weight | Evaluations scheduled at 7 days, 1 month, 3 months, 6 months and 12 months post embolization
  Weight loss expressed in percentage of total weight loss (%TWL)
Change in abdominal circumference | Evaluations scheduled at 1 month, 3 months, 6 months and 12 months post embolization
  Measurement of abdominal circumference in centimetres
Change in thigh circumferences | Evaluations scheduled at 1 month, 3 months, 6 months and 12 months post embolization
  Measurement of thigh circumferences in centimetres
Change in Ghrelinemia | Evaluations scheduled at 1 month, 3 months, 6 months and 12 months post embolization
  Measurement of serum ghrelin concentration
Change in Quality of life | Evaluations scheduled at 7 days, 1 month, 3 months, 6 months and 12 months post embolization
  Quality of Life is scored using Moorehead-Ardelt II Quality of life questionnaire. The questionnaire involves 6 questions scored from -0,5 to +0,5. The mean of the 6 answers leads to a sum between -3 (very poor quality of life) to +3 (very good quality of life).
Number of upper digestive endoscopies | 12 months after bariatric embolization
  Count of upper digestive endoscopies performed per patient during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Raoul POP, MD, PhD, Principal Investigator — Service de Neuroradiologie Interventionnelle, Nouvel Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Flegal KM. High body mass index for age among US children and adolescents, 2003-2006. JAMA. 2008 May 28;299(20):2401-5. doi: 10.1001/jama.299.20.2401. PMID 18505949
- [Background] Sturm R. Increases in morbid obesity in the USA: 2000-2005. Public Health. 2007 Jul;121(7):492-6. doi: 10.1016/j.puhe.2007.01.006. Epub 2007 Mar 30. PMID 17399752
- [Background] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982
- [Background] Baptista V, Wassef W. Bariatric procedures: an update on techniques, outcomes and complications. Curr Opin Gastroenterol. 2013 Nov;29(6):684-93. doi: 10.1097/MOG.0b013e3283651af2. PMID 24100715
- [Background] Aina R, Oliva VL, Therasse E, Perreault P, Bui BT, Dufresne MP, Soulez G. Arterial embolotherapy for upper gastrointestinal hemorrhage: outcome assessment. J Vasc Interv Radiol. 2001 Feb;12(2):195-200. doi: 10.1016/s1051-0443(07)61825-9. PMID 11265883
- [Background] De Wispelaere JF, De Ronde T, Trigaux JP, de Canniere L, De Geeter T. Duodenal ulcer hemorrhage treated by embolization: results in 28 patients. Acta Gastroenterol Belg. 2002 Jan-Mar;65(1):6-11. PMID 12014319
- [Background] Defreyne L, Vanlangenhove P, De Vos M, Pattyn P, Van Maele G, Decruyenaere J, Troisi R, Kunnen M. Embolization as a first approach with endoscopically unmanageable acute nonvariceal gastrointestinal hemorrhage. Radiology. 2001 Mar;218(3):739-48. doi: 10.1148/radiology.218.3.r01mr05739. PMID 11230648
- [Background] Goldman ML, LAND WC, Bradley EL, Anderson RT. Transcatheter therapeutic embolization in the management of massive upper gastrointestinal bleeding. Radiology. 1976 Sep;120(3):513-21. doi: 10.1148/120.3.513. PMID 1085008
- [Background] Holme JB, Nielsen DT, Funch-Jensen P, Mortensen FV. Transcatheter arterial embolization in patients with bleeding duodenal ulcer: an alternative to surgery. Acta Radiol. 2006 Apr;47(3):244-7. doi: 10.1080/02841850600550690. PMID 16613304
- [Background] Lang EV, Picus D, Marx MV, Hicks ME. Massive arterial hemorrhage from the stomach and lower esophagus: impact of embolotherapy on survival. Radiology. 1990 Oct;177(1):249-52. doi: 10.1148/radiology.177.1.2399325.
- [Background] Lieberman DA, Keller FS, Katon RM, Rosch J. Arterial embolization for massive upper gastrointestinal tract bleeding in poor surgical candidates. Gastroenterology. 1984 May;86(5 Pt 1):876-85. PMID 6608465
- [Background] Ljungdahl M, Eriksson LG, Nyman R, Gustavsson S. Arterial embolisation in management of massive bleeding from gastric and duodenal ulcers. Eur J Surg. 2002;168(7):384-90. doi: 10.1080/110241502320789050. PMID 12463427
- [Background] Miller M Jr, Smith TP. Angiographic diagnosis and endovascular management of nonvariceal gastrointestinal hemorrhage. Gastroenterol Clin North Am. 2005 Dec;34(4):735-52. doi: 10.1016/j.gtc.2005.09.001. PMID 16303580
- [Background] Morris DC, Nichols DM, Connell DG, Burhenne HJ. Embolization of the left gastric artery in the absence of angiographic extravasation. Cardiovasc Intervent Radiol. 1986;9(4):195-8. doi: 10.1007/BF02577940. PMID 3094950
- [Background] Ripoll C, Banares R, Beceiro I, Menchen P, Catalina MV, Echenagusia A, Turegano F. Comparison of transcatheter arterial embolization and surgery for treatment of bleeding peptic ulcer after endoscopic treatment failure. J Vasc Interv Radiol. 2004 May;15(5):447-50. doi: 10.1097/01.rvi.0000126813.89981.b6. PMID 15126653
- [Background] Rosch J, Dotter CT, Brown MJ. Selective arterial embolization. A new method for control of acute gastrointestinal bleeding. Radiology. 1972 Feb;102(2):303-6. doi: 10.1148/102.2.303. No abstract available. PMID 4536688
- [Background] Schenker MP, Duszak R Jr, Soulen MC, Smith KP, Baum RA, Cope C, Freiman DB, Roberts DA, Shlansky-Goldberg RD. Upper gastrointestinal hemorrhage and transcatheter embolotherapy: clinical and technical factors impacting success and survival. J Vasc Interv Radiol. 2001 Nov;12(11):1263-71. doi: 10.1016/s1051-0443(07)61549-8. PMID 11698624
- [Background] Toyoda H, Nakano S, Takeda I, Kumada T, Sugiyama K, Osada T, Kiriyama S, Suga T. Transcatheter arterial embolization for massive bleeding from duodenal ulcers not controlled by endoscopic hemostasis. Endoscopy. 1995 May;27(4):304-7. doi: 10.1055/s-2007-1005697. PMID 7555935
- [Background] Kipshidze N, Archvadze A, Bertog S, Leon MB, Sievert H. Endovascular Bariatrics: First in Humans Study of Gastric Artery Embolization for Weight Loss. JACC Cardiovasc Interv. 2015 Oct;8(12):1641-4. doi: 10.1016/j.jcin.2015.07.016. No abstract available. PMID 26493259
- [Background] Syed MI, Morar K, Shaikh A, Craig P, Khan O, Patel S, Khabiri H. Gastric Artery Embolization Trial for the Lessening of Appetite Nonsurgically (GET LEAN): Six-Month Preliminary Data. J Vasc Interv Radiol. 2016 Oct;27(10):1502-8. doi: 10.1016/j.jvir.2016.07.010. Epub 2016 Aug 24. PMID 27567998
- [Background] Weiss CR, Akinwande O, Paudel K, Cheskin LJ, Holly B, Hong K, Fischman AM, Patel RS, Shin EJ, Steele KE, Moran TH, Kaiser K, Park A, Shade DM, Kraitchman DL, Arepally A. Clinical Safety of Bariatric Arterial Embolization: Preliminary Results of the BEAT Obesity Trial. Radiology. 2017 May;283(2):598-608. doi: 10.1148/radiol.2016160914. Epub 2017 Feb 14. PMID 28195823
- [Background] Bai ZB, Qin YL, Deng G, Zhao GF, Zhong BY, Teng GJ. Bariatric Embolization of the Left Gastric Arteries for the Treatment of Obesity: 9-Month Data in 5 Patients. Obes Surg. 2018 Apr;28(4):907-915. doi: 10.1007/s11695-017-2979-9. PMID 29063494
- [Background] Pirlet C, Ruzsa Z, Costerousse O, Nemes B, Merkely B, Poirier P, Bertrand OF. Transradial left gastric artery embolization to treat severe obesity: A pilot study. Catheter Cardiovasc Interv. 2019 Feb 15;93(3):365-370. doi: 10.1002/ccd.27846. Epub 2018 Oct 4. PMID 30286527
- [Background] Elens S, Roger T, Elens M, Rommens J, Sarafidis A, Capelluto E, Delcour C. Gastric Embolization as Treatment for Overweight Patients; Efficacy and Safety. Cardiovasc Intervent Radiol. 2019 Apr;42(4):513-519. doi: 10.1007/s00270-018-2130-x. Epub 2018 Nov 28. PMID 30488305